CLINICAL TRIAL: NCT05572463
Title: A Randomized, Open-label, Multicenter, Multi-arm, Phase 1b/2 Platform Study to Evaluate Safety and Efficacy of Investigational Immunotherapies in Participants With Previously Treated Unresectable or Metastatic Melanoma
Brief Title: A Platform Study of Novel Immunotherapy Products in Participants With Previously Treated Unresectable or Metastatic Cutaneous Melanoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Strategy
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Collaborators: Innovent Biologics (USA), Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLATFORM201
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Unresectable Cutaneous Melanoma; Metastatic Cutaneous Melanoma
Keywords: Neoplasms; Melanoma; Malignant Melanoma
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — sintilimab

STUDY DESIGN:
Intervention Model Description: An open-label platform study that will allow evaluation of multiple novel IPs. The study will include multiple treatment arms that can be added sequentially or in parallel. There will be a master protocol describing study design elements common to all treatment arms with treatment arms described in the appendices, added through amendments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm 1 (Experimental): Sintilimab is a recombinant fully human anti-programmed cell death protein 1 (PD-1) monoclonal antibody, and IBI110 is a recombinant fully human anti-lymphocyte activation gene 3 (LAG3) monoclonal antibody. Sintilimab (IBI308) will be administered intravenously (IV) in combination with IBI110 administered intravenously (IV) every 3-weeks (Q3W).
  Interventions: Combination Product: Sintilimab + IBI110

INTERVENTIONS:
Combination Product: Sintilimab + IBI110 — IBI110 infusion in combination with Sintilimab (IBI308) infusion will be given on a Q3W schedule
  Other Names: Sintilimab (IBI308)

SUMMARY:
This is a platform study evaluating the safety and efficacy of multiple novel investigational products (IPs) that target unresectable or metastatic cutaneous melanoma in participants who have failed standard treatment.

DETAILED DESCRIPTION:
This is a Phase 1b/2, randomized, open label, multicenter, platform study evaluating the safety and efficacy of multiple novel investigational products (IPs) that target mechanisms implicated in resistance to immunotherapy in participants with unresectable or metastatic cutaneous melanoma who have resistance to anti-PD-1/L1 agents. This study will include multiple treatment arms that can be added sequentially or in parallel.

Each arm consists of a selection and expansion part. The selection part is used for evaluation of safety and preliminary efficacy in each arm. The selection part may also include a safety run-in portion for preliminary safety evaluation and dose confirmation prior to proceeding. If the criteria for safety and preliminary efficacy are met, the arm will open for additional enrollment in an expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, age 18 years or older
2. Histologically confirmed unresectable or metastatic cutaneous melanoma
3. Documented radiological progression on prior treatment(s) that included an anti-PD-1/L1 agent
4. Available tumor tissue OR be willing to provide a fresh tumor biopsy
5. Presence of at least one measurable lesion as assessed by CT and/or MRI according to RECIST 1.1
6. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1
7. Adequate organ and bone marrow function

Exclusion Criteria:

1. Known hypersensitivity to monoclonal antibodies, any of the IPs, or excipients contained in these products
2. Current anti-cancer therapy, other investigational treatment, or any participation in other interventional trials
3. Prior exposure to any therapy that targets the same target as the product under investigation, except for PD-1/L1
4. Known symptomatic/active untreated central nervous system (CNS) metastasis
5. Inadequate recovery from toxicity and/or complications attributable to any previous anti-cancer therapy
6. Inadequate recovery from all recent surgeries
7. At least 1-week from the time of minor surgery and at least 4 weeks from a major surgery
8. Received a live vaccine within 30 days prior to randomization (or planned to receive a live attenuated vaccine during the study)
9. History of HIV infection (positive HIV test, not on antiretroviral therapy, detectable viral load)
10. Active hepatitis B (positive hepatitis B surface antigen test) or hepatitis C infection (positive hepatitis C antibody)
11. Documented history or current diagnosis of clinically significant cardiac disease
12. History of or present CNS disease unrelated to cancer, unless adequately treated with standard medical therapy
13. Received solid organ or bone marrow transplantation
14. History of non-infectious pneumonitis requiring corticosteroid therapy within 1 year prior to enrollment, or current presence of interstitial lung disease
15. Active or previously documented autoimmune disease including but not limited to inflammatory bowel disease, diverticulitis, celiac disease, systemic lupus erythematosus, Wegener syndrome, multiple sclerosis, and vasculitis
16. Requiring long term systemic corticosteroids, except topical cortical steroids for intranasal inhalation or physiological dose
17. Active gastrointestinal (GI) bleeding or GI perforation or fistula
18. Serious active infection requiring intravenous (IV) antibiotics and/or hospitalization at study entry
19. Pregnant or lactating women or women who intend to get pregnant or lactate during the study and up to 120 days after the end of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability, and preliminary efficacy of novel immunotherapy IPs in participants with unresectable or metastatic melanoma that progressed while on prior treatment that included an anti-PD-1/L1 agent. (Selection Part) | Up to 28 months
  Incidence and severity of Adverse Events (AEs) and laboratory abnormalities
To evaluate the safety, tolerability, and preliminary efficacy of novel immunotherapy IPs in participants with unresectable or metastatic melanoma that progressed while on prior treatment that included an anti-PD-1/L1 agent. (Selection Part) | Day 1 to Day 42
  Incidence of dose-limiting toxicities (DLTs) [only applicable for safety run-in portion]
To identify novel immunotherapy IPs to progress into the expansion part (Selection Part) | Up to 2 years
  Overall response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
To evaluate the antitumor efficacy of immunotherapy in partcipants with unresectable or metastatic melanoma that progressed while on prior treatment(s) that included an anti-PD-1/L1 agent. (Expansion Part) | Up to 2 years
  ORR by RECIST 1.1

SECONDARY OUTCOMES:
To evaluate the preliminary anti-tumor efficacy by assessing additional endpoints of novel immunotherapy IPs (Selection Part) | Up to 4 years
  Duration of response (DOR) by RECIST 1.1
To evaluate the preliminary anti-tumor efficacy by assessing additional endpoints of novel immunotherapy IPs (Selection Part) | Up to 2 years
  Time to Response (TTR) by RECIST 1.1
To evaluate the preliminary anti-tumor efficacy by assessing additional endpoints of novel immunotherapy IPs (Selection Part) | Up to 2 years
  Disease control rate (DCR) by RECIST 1.1
To evaluate the preliminary anti-tumor efficacy by assessing additional endpoints of novel immunotherapy IPs (Selection Part) | Up to 4 years
  Progression-free survival (PFS) by RECIST 1.1
To evaluate the preliminary anti-tumor efficacy by assessing additional endpoints of novel immunotherapy IPs (Selection Part) | Up to 4 years
  Overall survival (OS)
To characterize the pharmacokinetic (PK) profile and immunogenicity (Selection, Expansion Part) | Up to 25 months
  Pharmacokinetic parameters including, but not limited to area under the concentration -time curve over dosing interval (AUCtau), Maximum observed plasma concentration at steady state (Cmax,ss), and trough plasma concentration at steady state (Ctrough,ss)
To characterize the pharmacokinetic (PK) profile and immunogenicity (Selection, Expansion Part) | Up to 25 months
  Prevalence and incidence of anti-product antibodies (ADA, Nab)
To evaluate anti-tumor efficacy by assessing additional endpoints by RECIST 1.1 (Expansion Part) | Up to 4 years
  Duration of response (DOR) by RECIST 1.1
To evaluate anti-tumor efficacy by assessing additional endpoints by RECIST 1.1 (Expansion Part) | Up to 2 years
  Time to Response (TTR) by RECIST 1.1
To evaluate anti-tumor efficacy by assessing additional endpoints by RECIST 1.1 (Expansion Part) | Up to 2 years
  Disease control rate (DCR) by RECIST 1.1
To evaluate anti-tumor efficacy by assessing additional endpoints by RECIST 1.1 (Expansion Part) | Up to 4 years
  Progression-free survival (PFS) by RECIST 1.1
To evaluate anti-tumor efficacy by assessing additional endpoints by RECIST 1.1 (Expansion Part) | Up to 4 years
  Overall survival (OS)
To further evaluate the safety and tolerability of novel immunotherapy IPs (Expansion Part) | Up to 28 months
  Incidence and severity of AEs and laboratory abnormalities

CONTACTS AND LOCATIONS:
Locations (13):
- United States (3):
  - University of California San Francisco Medical Center, San Francisco, California
  - Henry Ford Hospital, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
- Princess Victoria Hospital, Woolloongabba, Queensland, Australia
- France (2):
  - Hospices Civil De Lyon Nord - Centre Hospitalier Lyon Sud - Dermatologie, Lyon
  - Hospital Saint Louis, Paris
- Germany (2):
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Universitatsklinikum Essen, Essen
- Spain (2):
  - Institut Catala d'Oncologia Hospital Universitari Germans Trials I Pujol, Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Cordoba, Córdoba
- Universitaets Spital Zurich, Zurich, Switzerland
- United Kingdom (2):
  - Cambridge University Hospitals NHS Foundation Trust (Oxford), Cambridge
  - Lancashire Teaching Hospitals (Preston), Preston